CLINICAL TRIAL: NCT04146090
Title: Low-pressure vs Standard-pressure in Laparoscopic Cholecystectomy. A Randomized Controlled Trial Evaluating the Quality of Recovery Measured by QoR-40
Brief Title: Low-pressure vs Standard-pressure in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Toshiyuki Moro, Professor, Pontificia Universidade Catolica de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CAAE 18245019.6.0000.5373
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2019-10

CONDITIONS: Laparoscopic Surgery; Pneumoperitoneum; Cholecystitis; Choledocholithiasis; Quality of Life; Postoperative Nausea and Vomiting; Postoperative Pain; Satisfaction, Patient
MeSH Terms: conditions — Pneumoperitoneum; Cholecystitis; Choledocholithiasis; Postoperative Nausea and Vomiting; Pain, Postoperative; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Double blinded, randomised controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomised in a 1:1 ratio (www.random.org) into 2 groups: LP (low-pressure) or S (standard). Group assignments will be sealed in sequentially numbered opaque envelopes that will be opened after patient inclusion into the study. Care providers, researchers, and patients will be blinded to group assignments.Insufflation pressure will be maintained in 14 mmHg (group S) or 10 mmHg (group LP). Anesthesiologists and surgeons will not have access to insufflation pressure display (it will be covered by an opaque paper and will be set by operating room personnel).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-pressure (Active Comparator): Forty patients aged 18 to 65 years, with an ASA physical status I or II, who will be scheduled to undergo laparoscopic cholecystectomy
  Interventions: Other: Low-pressure pneumoperitoneum
- Standard pressure (Placebo Comparator): Forty patients aged 18 to 65 years, with an ASA physical status I or II, who will be scheduled to undergo laparoscopic cholecystectomy
  Interventions: Other: Standard pressure pneumoperitoneum

INTERVENTIONS:
Other: Low-pressure pneumoperitoneum — Pneumoperitoneum will be maintained in 10 mmHg
  Arms: Low-pressure
Other: Standard pressure pneumoperitoneum — Pneumoperitoneum will be maintained in 14 mmHg
  Arms: Standard pressure

SUMMARY:
Background. Many studies have demonstrated reduced postoperative pain in patients undergoing lower pneumoperitoneum pressure level during laparoscopic cholecystectomy. However, most of them has shown a high risk of bias and low or very low quality of evidence. Considering the need to evaluate, not only the postoperative pain, but the effect of anesthesia and surgery on patient recovery and satisfaction, we have designed a prospective, randomised and double-blinded study to evaluate the quality of recovery, using the Quality of Recovery Questionnaire (QoR-40), in patients undergoing LC under low-pressure or standard pressure pneumoperitoneum. Methods. Eighty patients aged 18 to 65 years of age will be randomised into 2 groups: LP (low-pressure - 10mmHg) or S (standard - 14 mmHg) enrolled in the study. Anesthesia will be induced with remifentanil, propofol and rocuronium and the maintenance will be achieved with sevoflurane and remifentanil Anesthesiologists and surgeons will not have access to insufflation pressure display. The primary outcome will be assessed using the Quality of Recovery Questionnaire (QoR-40) which is a 40-item quality of recovery scoring system. In addition, the intraoperative rocuronium consumption, time to eye opening (time from the discontinuation of anesthetics to eye opening), post-operative nausea and vomiting, pain score, analgesic use, and length of PACU stay (time to Aldrete score ≥ 9) will be recorded.

DETAILED DESCRIPTION:
INTRODUCTION

Laparoscopic cholecystectomy (LC) is currently one of the most commonly performed surgical procedures worldwide. Although it is generally a procedure of short duration and a growing number of patients are being treated on an outpatient basis, post-operative pain remains a major reason for prolonged hospital stay, and readmission.1 A number of trials have evaluated methods to prevent postoperative pain after LC. One of the most tested was low-pressure pneumoperitoneum (7-10 mmHg) when compared to standard-pressure (12-16 mmHg).2-10 It is well known that carbon dioxide pneumoperitoneum provides adequate working space and organ visualization but this may cause several physiologic changes. Many studies have demonstrated reduced postoperative pain in patients undergoing lower pneumoperitoneum pressure level. However, a recent Cochrane systematic review have shown a high risk of bias and low or very low quality of evidence in 20 trials from 21 evaluated. Additionally, the decrease in the effective working space provided by lower intra-abdominal pressure may increase the technical difficulty, the incidence the procedure-related injuries and the operative time. 11 Considering the measurements that assess quality of life from the patient's perspective are increasingly recognized as an important quality metric in perioperative clinical trials, and the need to evaluate, not only the postoperative pain, but the effect of anesthesia and surgery on patient recovery and satisfaction, we have designed a prospective, randomised and double-blinded study to evaluate the quality of recovery, using the Quality of Recovery Questionnaire (QoR-40) 12, in patients undergoing LC under low-pressure or standard pressure pneumoperitoneum. Additionally, clinical variables, including time to eye opening, procedural time, cumulative dose of rocuronium, conversion to open surgery, surgeons' satisfaction, the occurrence of nausea and vomiting, pain score, use of analgesics, and length of Post Anesthetic Care Unit (PACU) stay was determined.

METHODS

Study Population This randomised trial was approved by the Research Ethics Committee of the School of Medical and Health Sciences, Pontifical Catholic University of São Paulo (Sorocaba, São Paulo - Brazil), on 13 August 2019, 18245019.6.0000.5373 (Chairperson Prof. J.A. Costa). Written informed consent will be obtained from all participants. Eighty patients aged 18 to 65 years of age, with an AmericanSociety of Anesthesiologists (ASA) physical status I or II, who will be scheduled to undergo LC at Santa Lucida Hospital, will be enrolled in the study. Exclusion criteria prior to randomization will include: (i) refusal to participate; (ii) altered level of consciousness or inability to communicate; (iii) presented with a contraindication to any of the drugs used in the present study; (iv) history of alcohol or drug abuse; (v) a body mass index (BMI) ≥ 40; (vi) presence of chronic pain or using opioid; (vii) history of complicated gallstone diseases like acute cholecystitis, cholangitis or pancreatitis. Reasons for exclusion following randomization will include; (i) protocol violations, such as the use of medications not contemplated in the study protocol; (ii) conversion to an open surgical technique. Subjects will be randomised in a 1:1 ratio (www.random.org) into 2 groups: LP (low-pressure) or S (standard). Group assignments will be sealed in sequentially numbered opaque envelopes that will be opened after patient inclusion into the study. All care providers, researchers, and patients will be blinded to group assignments.

Anesthetic and Surgical Management Premedication will not be administered. Patients will arrive at operation room (OR) after an 8-hour fast. Standard ASA monitors will be applied upon entry into the operating room and anesthesia will be induced with remifentanil 0.5 mcg. kg-1.min-1 over 3 min followed by propofol 2.0 mg.kg-1 and rocuronium 0.6 mg.kg-1 before tracheal intubation. Anesthetic maintenance will be achieved with sevoflurane 1% - 3% and remifentanil 0.3 mcg.kg-1min-1 whenever necessary to keep mean arterial pressure (MAP) and heart hate (HR) within ± 20% baseline values. Ventilation will be controlled mechanically to maintain an end-tidal carbon dioxide concentration of 30-40 mmHg. Oxygen and air will be administered in a ratio of 50%. Insufflation pressure will be maintained in 14 mmHg (group S) or 10 mmHg (group LP). Anesthesiologists and surgeons will not have access to insufflation pressure display (it will be covered by an opaque paper and will be set by operating room personnel). Patients who exhibited reductions in systolic arterial pressure (SAP) greater than 30% will be given ephedrine (10 mg). Normal saline will be used for fluid replacement therapy at a rate of 500 mL throughout the first 30 minutes, and, then, 2 mL.kg-1.h-1 until the end of the surgical procedure. All participants will be given dexamethasone (8 mg) and ketoprofen (100 mg) at the onset of surgery and ondansetron (4 mg) 15 minutes prior the end of the procedure. Atropine (0.01 mg. kg-1) and neostigmine (0.015 mg. kg-1) will be used to achieve T4/T1>0.9 on the Train-of-four (TOF) monitor prior to extubation. At the end of surgery, intra-abdominal irrigation with normal saline will be performed and the pneumoperitoneum will be carefully evacuated by manual compression. A total of 20 mL ropivacaine 0.75% will be injected to the subcutaneous tissue, fascia and parietal peritoneum through the port sites by the surgeon. The surgical working conditions will be scored according to an ordinal scale ranging from 1 (extremely poor conditions), 2 (poor conditions), 3 (acceptable conditions), 4 (good conditions) and 5 (optimal conditions). 13 All surgical procedures will be performed by the same team composed of three experienced surgeons.

The primary outcome will be assessed using the Quality of Recovery Questionnaire (QoR-40) which is a 40-item quality of recovery scoring system. In addition, the intraoperative rocuronium consumption, time to eye opening (time from the discontinuation of anesthetics to eye opening), post-operative nausea and vomiting, pain score, analgesic use, and length of PACU stay (time to Aldrete score ≥ 9) will be recorded. Pain will be assessed (at rest and after asking to cough) using a 0-10 numeric pain rating scale (NRS), where zero means no pain and 10 the worst imaginable pain. Analgesia will be provided with IV morphine every 5 minutes to maintain a pain score below 4 (2 mg when the pain score was <7 and 3 mg when it was ≥7). Following discharge from the PACU (minimum stay 60 minutes and Aldrete score ≥ 9), all of the participants will be given IV ketoprofen (100 mg) every 12 hours and oral dipyrone every six hours. Whenever patients judge their analgesia to be insufficient, oral tramadol (100 mg) will be administered at eight-hour minimum intervals. Postoperative nausea and vomiting (PONV) will be treated with dimenhydrinate (30 mg) intravenously. An investigator who will be blinded to group assignment will collect all postoperative outcome data 24 hours following the surgical procedure. The severity of pain was measured at 15-min intervals during PACU stay and at 4, 6, and 24 h after surgery. Tramadol consumption and the occurrence of nausea and vomiting episodes will be also recorded. These findings will be confirmed with the ward nursing staff. All study patients will be admitted to the hospital for a minimum of 24 hours.

Data Collection The baseline QoR-40 questionnaire will be provided to subjects after informed consent is obtained in the preoperative holding area, 12 hours after surgery and in the next day by a blinded investigator. The QoR-40 questionnaire assesses five dimensions of recovery (physical comfort - 12 items; emotional state - 7 items; physical independence - 5 items; physiological support - 7 items; and pain - 7 items). Each item was rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR-40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).

Statistical Analysis The sample size will be calculated considering 90% power to detect a 10-point difference in QoR-40, which indicates the need to include 31 participants in each group.

A 10-point difference represents a 15% improvement in the quality of recovery on the basis of previously reported values of the QoR-40.12,14 Taking possible losses into consideration, the final sample will include 80 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ASA physical status I or II, who will be scheduled to undergo LC

Exclusion Criteria:

* (i) refusal to participate; (ii) altered level of consciousness or inability to communicate; (iii) presented with a contraindication to any of the drugs used in the present study; (iv) history of alcohol or drug abuse; (v) a body mass index (BMI) ≥ 40; (vi) presence of chronic pain or using opioid; (vii) history of complicated gallstone diseases like acute cholecystiitis, cholangitis or pancreatitis. Reasons for exclusion following randomization will include; (i) protocol violations, such as the use of medications not contemplated in the study protocol; (ii) conversion to an open surgical technique

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Quality of recovery | 24 hours after surgery
  The primary outcome will be assessed using the Quality of Recovery Questionnaire (QoR-40) which is a 40-item quality of recovery scoring system

SECONDARY OUTCOMES:
Postoperative pain | The severity of pain was measured at 15-min intervals during PACU stay and at 4, 6, and 24 hours after surgery
  Pain will be assessed (at rest and after asking to cough) using a 0-10 numeric pain rating scale (NRS), where zero means no pain and 10 the worst imaginable pain.
Postoperative nausea and vomiting | 24 hours
  Occurrence of nausea and vomiting
Intraoperative rocuronium consumption | Intraoperative
  Rocuronium consumption in mg/kg
Time to eye opening | Intraoperative (During recovery in operation room)
  Time from the discontinuation of anesthetics to eye opening
Surgical working conditions | Intraoperative
  Surgeon will score surgical conditions according to an ordinal scale ranging from 1 (extremely poor conditions), 2 (poor conditions), 3 (acceptable conditions), 4 (good conditions) and 5 (optimal conditions)

CONTACTS AND LOCATIONS:
Locations (1):
- Eduardo T Moro, Araçoiaba da Serra, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No